CLINICAL TRIAL: NCT03946020
Title: Bovine Derived Xenograft in Combination With Autogenous Bone Chips Versus Xenograft Alone for the Augmentation of Bony Dehiscences Around Oral Implants: a Randomized, Controlled, Split-mouth Clinical Trial
Brief Title: GBR and Autogenous Bone Chips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Wim Teughels, Clinical Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S55609
Record Dates: First submitted 2019-05-02; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Bone Resorption
Keywords: implants; GBR; DBBM; grafts; bone
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Split mouth
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmentation with autologous bone + DBBM (Active Comparator): A layer of autogenous bone chips was placed on the implant surface. On top of this a layer of DBBM (Bio-Oss™, Geistlich®, Wolhusen, Switserland) was placed, thereafter covered with a collagen membrane.
  Interventions: Procedure: Guided bone regeneration with or without autologous bone
- Augmentation with DBBM (Experimental): A layer of DBBM was placed on the implant surface and thereafter covered with a collagen membrane. Care was taken to make both augmentations as comparable as possible by weighting the used amount of graft material.
  Interventions: Procedure: Guided bone regeneration with or without autologous bone

INTERVENTIONS:
Procedure: Guided bone regeneration with or without autologous bone — Autogenous bone chips were collected. On each side a bone level implant was placed. The bone dehiscence was measured and was thereafter treated according to the GBR protocol. A resorbable native collagen was adapted to the defect.

SUMMARY:
This study will be an open, prospective, split-mouth, randomised controlled clinical trial. A total of 14 patients searching for oral implant treatment and where a GBR procedure is indicated per implant treatment will be enrolled.

All patients have to fulfill all of the inclusion criteria and none of the exclusion criteria. From all patients clinical photos will be taken.

Two sites within a patient will be randomly allocated to the 'autologous bone chips and DBBM or 'DBBM particles alone' group.

The study will be 1 year follow-up study comprising 9 visits

DETAILED DESCRIPTION:
A randomized controlled clinical trial (RCT) to compare the use of deproteinized bovine bone mineral (DBBM) in combination with autogenous bone chips versus a DBBM alone for the augmentation of bony dehiscence after dental implant placement

Objectives: 1. To test whether the use of DBBM is not inferior to the use of a combination of DBBM and autogenous bone chips for the filling of bony dehiscence around dental implants

2. To test whether a digital impression technique can be used to measure guided bone regeneration in comparison to conventional measurement with a dental probe and to compare these observations with cone beam CT images

Study Design: Randomized, controlled, single center, split mouth study

Study Population: Partially edentulous male or female patients in need for oral implants for a fixed prosthetic implant supported rehabilitation and where a Guide Bone Regeneration (GBR) procedure is indicated during implant treatment

Patient Number: 14

Duration of treatment: The time in the study for each patient will be 1 year and 4 months. The treatment period includes implant and abutment installation (in a twostage procedure), with a healing time of minimum 12 weeks before the start of the prosthetic phase.

Study devices: Implants: 3.3 / 4.1 / 4.8 mm Straumann Bone level implants Bone Graft: DBB (Demineralised Bovine Bone, Bio OSS) Measuring Devices: Cadent iTero & software and Dental Probes Prosthetics: Straumann (computer aided design computer aided manufacturing (CAD CAM) crowns and abutments

Outcome variables:

Primary outcome variable: Difference in bone fill between DBB + bone chips vs. DBB without bone chips afer 24 weeks of submerged healing. The "ideal bone volume" as defined at base line (= 100%) will be compared to the received bone fill [%] at re-entry measured by a digital impression technique (before and after GBR, and at abutment connection, before and after raising a flap, and at the 1-year follow-up).

The method of digital impression will be compared to CBCT immediately after implant placemetn and 1 year and periodontal probing during surgery and re-enty

Secondary Parameters:

Page 5 of 35 A comparison of 3 different tools (probe, CBCT and digital impression) for measuring the bone volume changes in relation to GBR procedures. Implant survival en success rates on a patient and implant level Marginal bone level alterations

Safety: Adverse Events / Adverse Device Effects

ELIGIBILITY:
Inclusion Criteria:

* > 18 years,
* in need of a solitary implant in quadrant 1 and 2 or quadrant 3 and 4 with simultaneous GBR procedure
* presence of a pre-operative CBCT.

Exclusion Criteria:

* smokers
* patients with systemic diseases that could interfere with the healing
* patients undergoing bisphosphonate treatment
* patients who previously received radiation therapy of the jaws
* patients that received a GBR procedure in the region of interest in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Horizontal and vertical bone augmentation | 16 weeks
  The change of dimension was assessed comparing Cone Beam Computed Tomography scans (CBCT)

SECONDARY OUTCOMES:
Success of grafting procedure as assessed by clinical interpretation | 1 year
  Defined as no persistent pain in the grafted area and no suppuration or expulsion of graft material and implant survival rates being lack of mobility, absence of peri-implant radiolucency, absence of recurrent peri-implant infection with suppuration, absence of continuous or recurrent pain, and no structural failure of the implant
Marginal bone level alterations assessed on peri-apical radiographs using software (ImageJ) | 1 year
  measured from a reference point (implant shoulder) to the most coronal point of BIC, both mesially and distally

CONTACTS AND LOCATIONS:
Overall Officials: Andy Temmerman, DDS, MSc, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Temmerman A, Cortellini S, Van Dessel J, De Greef A, Jacobs R, Dhondt R, Teughels W, Quirynen M. Bovine-derived xenograft in combination with autogenous bone chips versus xenograft alone for the augmentation of bony dehiscences around oral implants: A randomized, controlled, split-mouth clinical trial. J Clin Periodontol. 2020 Jan;47(1):110-119. doi: 10.1111/jcpe.13209. Epub 2019 Nov 5. PMID 31602699